CLINICAL TRIAL: NCT05479201
Title: Prevalence of Obstructive Sleep Apnoea (OSA) Among 4-8 Years Old Children in the General Population
Status: Completed | Type: Observational
Sponsor: Akureyri Hospital (Other Government)
Collaborators: MyCardio (Unknown)
Responsible Party: Sponsor
Other Study IDs: VSN-22-096
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children 4-8 years of age
  Interventions: Diagnostic Test: Home based sleep test

INTERVENTIONS:
Diagnostic Test: Home based sleep test — Home based sleep test to calculate apnea hypopnea index (AHI) for evaluation of sleep apnea, sleep quality (SQI) and sleep duration (SD)
  Other Names: SleepImage (FDA K182618)

SUMMARY:
The purpose of this study is to estimated prevalence of obstructive sleep apnea (OSA) in 4-8 year old children. To date, most studies estimating prevalence of sleep apnea in young children are based on utilizing subjective questionnaires. The few studies that have utilized objective sleep measures have tested only those children suspected of sleep apnea based on subjective questionnaires, finding prevalence in the range of 1-13%. Untreated OSA is associated with significant morbidities in children, affecting their behavior, cognitive development, cardiovascular-and cardio metabolic health, endocrine and immune function. Better understanding of prevalence of sleep apnea in young children should be beneficial. This study will help to understand the prevalence of sleep apnea in each age-group of children 4-8 years of age and whether certain groups, such as children with obesity or asthma have higher prevalence and/or more severe disease.

The primary objective of this study is to get better understanding of prevalence and severity of sleep apnea in young children using objective sleep measures for all participants.

DETAILED DESCRIPTION:
The study is a population-based, observational study of 4-8 year old children located in Akureyri, Iceland. All parents in this geographical area will be invited for their child/children to participate in the study.

Parents of all participating children will be asked to answer questionnaires to assess general health, sleep habits, behavior and quality of life and then measure their sleep for five consecutive nights with a home based sleep test.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-8-years old

Exclusion Criteria:

* Children with atrial fibrillation or ventricular trigemini

Ages: 4 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: All children in a pre-specified geographical area 4-8 years of age
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA in 4-8 year old children | Baseline
  Apnea Hypopnea Index (AHI)

SECONDARY OUTCOMES:
Prevalence of OSA defined by a specific age range (4-5-year-old/5-6-year-old/6-7-year-old/7-8-year-old) | Baseline
  Apnea Hypopnea Index (AHI)

OTHER OUTCOMES:
Intra-night variability in OSA | Baseline
  Apnea Hypopnea Index (AHI)

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Pedersen, MD, Principal Investigator — University of Iceland
Locations (1):
- Sjukrahusid a Akureyri, Akureyri, Iceland

IPD SHARING:
Plan to Share IPD: No